CLINICAL TRIAL: NCT06409325
Title: Effectiveness of Magnetic Seizure Therapy Versus Electroconvulsive Therapy for Major Depressive Episode
Brief Title: Effectiveness of MST Versus ECT for Major Depressive Episode
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Tianhong ZHANG, Associate Professor, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NS70002024
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Electroconvulsive therapy (ECT); magnetic seizure therapy (MST)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The present clinical protocol is designed as a double-blind, parallel, non-inferiority, randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both clinical staff and participants were blinded to the treatment assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the MST group (Experimental): MST was conducted at 100 Hz and 100% output using a pulse width of 350 μs and a peak intensity of the magnetic field at 3.0 Tesla. The duration of magnetic stimulation was titrated using a 10-second train duration, starting from 2 seconds and increasing by 4 seconds in subsequent sessions, up to a maximum of 10 seconds (i.e., 200-1,000 pulses per session). In cases of poor seizure quality (<15 s), the stimulation duration increment was set to 6 seconds in the next session. If no seizures were elicited, an additional 10-second stimulation was administered immediately. Subsequent MST treatments were maintained at a 10-second duration for a total of 1000 pulses.
  Interventions: Device: MST
- the ECT group (Active Comparator): For ECT, the pulse width of the electrical stimulus was set to 0.5 ms. The initial energy dosage was determined based on the patient's age, with subsequent sessions increasing by 5% increments. In cases of inadequate seizure duration (<25 s), the maximum dosage was administered in the following session. If no seizures were induced, the maximum dosage was administered immediately.
  Interventions: Device: ECT

INTERVENTIONS:
Device: MST — MST was delivered with NS 7000 (Wuhan Yiruide Medical Equipment New Technology Co., Ltd.) using a round coil (125-mm diameter) positioned on the vertex.
  Arms: the MST group
Device: ECT — The bitemporal ECT procedure utilized the Thymatron System IV device (Somatics, USA).
  Arms: the ECT group

SUMMARY:
Despite advancements in Magnetic Seizure Therapy (MST) and Electroconvulsive Therapy (ECT) for Major Depressive Disorder (MDD), there remains a need for further research to replicate clinical outcomes and understand the therapeutic targets of these treatments. This study aims to address these gaps through a double-blinded, randomized, non-inferiority investigation comparing the efficacy, tolerability, cognitive adverse effects, and neurophysiological biomarkers of MST and bilateral ECT in patients with MDD.

DETAILED DESCRIPTION:
Participants will be randomly allocated to either the ECT or MST group. Each center aims to recruit 30 participants for each group, using block randomization, resulting in a total of 30 participants per group. The trial comprises a 12-session intervention phase of ECT/MST, spanning approximately 4 weeks, followed by a 12-week observation period. For the first three treatment sessions, participants will receive consecutive sessions. Subsequently, there will be a one-day interval between sessions 4 to 6, a two-day interval between sessions 7 to 9, and a three-day interval between sessions 10 to 12, ensuring completion within a month. Following treatment completion, participants will undergo follow-up clinical observations every four weeks for 12 weeks. EEG and ECG recordings will be obtained at baseline, post-session 3, 6, 9, 12 (3 hours after each session), and at the 12-week follow-up. All evaluations will be conducted under standardized conditions throughout the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the diagnostic criteria for MDD as outlined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
* Participants must have a baseline score of 18 or higher on the 24-item Hamilton Depression Rating Scale (HDRS-24).
* During the trial's treatment period, participants must be using a single antidepressant medication at a stable dose.
* Participants must be between the ages of 18 and 65 years.
* Informed consent from both parents and legal guardians is required.

Exclusion Criteria:

* Individuals with current or history of organic brain disorders or neurological disorders will be excluded from the study.
* Participants with a Wechsler Abbreviated Scale of Intelligence (WASI) score of less than 70 will be excluded.
* Individuals currently taking antiepileptic drugs, benzodiazepines, or other medications that may affect seizure activity will be excluded from the study.
* Those with exposure to ECT, modified ECT, MST, transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), or other neurostimulation treatments in last 6 months will be excluded.
* Individuals with cochlear implants, cardiac pacemakers, implanted devices, or metal in the brain will be excluded from participation.
* Pregnant or lactating individuals will be excluded from the study.
* Individuals currently participating in another concurrent clinical trial will not be eligible for inclusion.
* Participants who refuse to provide informed consent to participate in the trial will be excluded.
* Other circumstances deemed unsuitable for participation by researchers will result in exclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
the response rate | 12 weeks
  It will be determined by Hamilton Depression Scale(HAMD-24 item) score. Specifically, the response rate is defined as a reduction of at least 50% in the HDRS-24 score from baseline.
the remission rate | 12 weeks
  It will be determined by Hamilton Depression Scale(HAMD-24 item) score. Specifically, the remission rate is defined as a reduction of at least 60% in the HDRS-24 score and a total score of 8 or less.

CONTACTS AND LOCATIONS:
Overall Officials: TianHong Zhang, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang T, He Y, Liu S, Ju M, Yang Y, Zhou R, Hong Y, Wei Y, Tang X, Zheng H, Jia Y, Liu H, Zhou D, Hu Q, Wang R, Zheng W, Zeng L, An C, Li C, Wang J. Effectiveness of magnetic seizure therapy versus electroconvulsive therapy for major depressive episode in China: protocol for a double-blind, randomized, non-inferiority trial. Front Psychiatry. 2025 Oct 23;16:1657906. doi: 10.3389/fpsyt.2025.1657906. eCollection 2025. PMID 41210143